CLINICAL TRIAL: NCT00716846
Title: Effects of Three Statins, Simvastatin, Atorvastatin, and Pitavastatin, on the Pharmacokinetics for Midazolam in Healthy Volunteers
Brief Title: Effects of Statins on the Pharmacokinetics for Midazolam in Healthy Volunteers
Acronym: H-17-21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Naoki Inui, Clinical Pharmacology and Therapeutics, Hamamatsu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Hamamatsu 18-21
Record Dates: First submitted 2008-07-10; First posted 2008-07-16 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2009-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Simvastatin; Atorvastatin; pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- statin-1 (Active Comparator): simvastatin
  Interventions: Drug: simvastatin
- statin-2 (Active Comparator): atorvastatin
  Interventions: Drug: atorvastatin
- statin-3 (Active Comparator): pitavastatin
  Interventions: Drug: pitavastatin

INTERVENTIONS:
Drug: simvastatin — 10mg, 2 weeks
  Other Names: Lipovas tablets
  Arms: statin-1
Drug: atorvastatin — 10mg
  Other Names: Lipitor tablets
  Arms: statin-2
Drug: pitavastatin — 2mg
  Other Names: Livalo tablets
  Arms: statin-3

SUMMARY:
The purpose of this study is to investigate whether statins have any influence on cytochrome P450 (CYP) 3A4 enzyme activity using a probe drug midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers in good health according to their medical history, a physical examination and standard laboratory tests

Exclusion Criteria:

* Subjects who have been using any continuous medication or herbal supplements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
the pharmacokinetics of oral midazolam | after 14-days treatment with statins

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Watanabe, MD,PhD, Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan